CLINICAL TRIAL: NCT04853992
Title: Phase 2a Trial to Assess the Efficacy and Safety of LEO 152020 in Adult Patients With Cholinergic Urticaria
Brief Title: Trial to Assess the Efficacy and Safety of LEO 152020 in Adult Patients With Cholinergic Urticaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EXP-2177; 2020-004961-38 (EudraCT Number)
Record Dates: First submitted 2021-04-20; First posted 2021-04-22 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Cholinergic Urticaria

STUDY DESIGN:
Intervention Model Description: Each treatment period will last 7 days with a wash-out period of 7 days between treatments
Who Masked: Participant, Investigator
Masking Description: Placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active - Placebo (Experimental): Patients will receive active treatment for 7 days, followed by a washout period of 7 days and then placebo for 7 days
  Interventions: Drug: LEO 152020; Drug: LEO 152020 placebo
- Placebo - Active (Experimental): Patients will receive placebo for 7 days, followed by a washout period of 7 days and then active treatment for 7 days
  Interventions: Drug: LEO 152020; Drug: LEO 152020 placebo

INTERVENTIONS:
Drug: LEO 152020 — LEO 152020 is a small drug molecule which can block the histamine 4 receptor (H4R). LEO 152020 is a tablet for oral administration.
Drug: LEO 152020 placebo — LEO 152020 placebo is a tablet for oral administration. LEO 152020 placebo contains the same excipients in the same concentration as the LEO 152020 tablet, except the medical ingredient, LEO 152020.

SUMMARY:
Phase 2a trial to assess the efficacy and safety of LEO 152020 in adult patients with cholinergic urticaria

DETAILED DESCRIPTION:
This is a phase 2a, randomised, double-blind, placebo-controlled, cross-over trial conducted in Germany at 3-6 sites. Subjects will be randomised to one of two treatment sequences (A and B). Each treatment period will last 7 days with a wash-out period of 7 days between treatments. Half of the subjects will start with treatment A followed by treatment B while the other half will start with treatment B followed by treatment A. A safety follow-up visit will be performed 3 days after last dose of the tested medication.

The main assessment is an urticaria activity score. After a Pulse-controlled ergometry (PCE) provocation test subjects will be rated on their number of wheals and their itch severity, resulting in a sum score ranging from 0 to 6 points.

ELIGIBILITY:
Main Inclusion Criteria:

* Subject with a history of Cholinergic urticaria diagnosis for ≥ 6 months
* Subject has active and uncontrolled Cholinergic urticaria disease at the time of screening and randomisation, as defined by the following:

  1. Urticaria control test < 12 at screening
  2. Urticaria Activity Score post-provocation ≥ 3
* Recent history (within 6 months of screening) with documented inadequate response to standard dose as to marketing authorization of H1 antihistamines.

Main Exclusion Criteria:

* Other clearly dominating forms* of urticaria as aetiology for wheal and flare type reactions

  *These diseases are allowed as comorbidities, if cholinergic urticaria is the dominating form of chronic urticaria,
* Systemic immunosuppressive medications within 4 weeks prior to screening,
* Systemic drugs (e.g. oral drug) with antihistamine properties including H1 antihistamines and some antidepressants (e.g. tricyclic antidepressants) and H2 antihistamines 1 week prior to randomisation and throughout the trial. However, topical antihistamines in the form of nasal spray and eyedrops are allowed in the standard prescribed dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (6):
- Germany (6):
  - LEO Investigational Site, Aachen
  - LEO Investigational Site, Berlin
  - LEO Investigational Site, Dresden
  - LEO Investigational Site, Freiburg im Breisgau
  - LEO Investigational Site, Kiel
  - LEO Investigational Site, München

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Access Criteria: De-identified Individual Participant Data can be made available to researchers and is subject to approved scientifically sound research proposal and signed data-sharing agreement.
URL: https://www.leopharmatrials.com/en/for-professionals

REFERENCES:
- [Derived] Grekowitz E, Metz M, Altrichter S, Bauer A, Brockow K, Heine G, Lionnet L, Saday KK, Hultsch T, Soerensen OE, Maurer M. Targeting histamine receptor 4 in cholinergic urticaria with izuforant (LEO 152020): results from a phase IIa randomized double-blind placebo-controlled multicentre crossover trial. Br J Dermatol. 2024 May 17;190(6):825-835. doi: 10.1093/bjd/ljae038. PMID 38308655

RESULTS

PARTICIPANT FLOW:
Groups:
- Active - Placebo: Patients will receive active treatment for 7 days, followed by a washout period of 7 days and then placebo for 7 days
  LEO 152020: LEO 152020 is a small drug molecule which can bind to the histamine 4 receptor (H4R). LEO 152020 is a tablet for oral administration.
  LEO 152020 placebo: LEO 152020 placebo is a tablet for oral administration. LEO 152020 placebo contains the same excipients in the same concentration as the LEO 152020 tablet, except the medical ingredient, LEO 152020.
- Placebo - Active: Patients will receive placebo for 7 days, followed by a washout period of 7 days and then active treatment for 7 days
  LEO 152020: LEO 152020 is a small drug molecule which can bind to the histamine 4 receptor (H4R). LEO 152020 is a tablet for oral administration.
  LEO 152020 placebo: LEO 152020 placebo is a tablet for oral administration. LEO 152020 placebo contains the same excipients in the same concentration as the LEO 152020 tablet, except the medical ingredient, LEO 152020.
Period: Treatment Period A
Arm/Group | Active - Placebo | Placebo - Active
Started | 11 | 9
Completed | 11 | 8
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Wash Out
Arm/Group | Active - Placebo | Placebo - Active
Started | 11 | 8
Completed | 10 | 8
Not Completed | 1 | 0
Not completed — Met exclusion criteria for next treatment phase | 1 | 0
Period: Treatment Period B
Arm/Group | Active - Placebo | Placebo - Active
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active - Placebo | Placebo - Active | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Median (Full Range); unit: years] | 25 [22 to 56] | 25 [20 to 47] | 25 [20 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 8 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Post-provocation Urticaria Activity Score (UASprovo)
Description: The Urticaria Activity Score (UAS) rates a participants' number of wheals and their itch severity on a scale from 0 to 6, with 6 being the most severe. UAS is assessed after provocation of urticaria by moderate exercise to cause sweating.
Time Frame: Baseline to Day 7
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Active: In this cross over study all participants received active treatment.
- Placebo: In this cross over study all participants received placebo
Arm/Group | Active | Placebo
Number analyzed (Participants) | 19 | 18
scores on a scale | -1.1 (2.1) | -0.5 (1.7)
Statistical Analysis 1: Comparison: Active vs Placebo; The primary endpoint, change from baseline in post-provocation Urticaria Activity Score (UASprovo) to the end of the treatment period, was compared between treatments with the null hypothesis that they are equal against the alternative that they are different. The primary efficacy endpoint was analysed using a linear mixed model, containing treatment, period and carryover effects, the factor site and additionally the value of UASprovo at baseline as a covariate; Test type: Superiority; p = 0.277, Mixed Models Analysis; Mean Difference (Net) = -0.58, 95% CI 2-sided [-1.69 to 0.53], Standard Error of Mean 0.5

2. Secondary Outcome: Number of Treatment Emergent Adverse Events
Time Frame: From start of each treatment period (day 1 for the 1st treatment period or day 15 or 22 for the 2nd treatment period) until 3 days after end of each treatment period (day 11 for the 1st treatment period or day 25 or 32 for the 2nd treatment period)
Population: Safety analysis set
Measure: Number; unit: Number of AEs
Arm/Group | Active | Placebo
Number analyzed (Participants) | 19 | 19
Number of AEs | 9 | 5

ADVERSE EVENTS:
Time Frame: From first trial related activity (up to 21 days before day 1 in first treatment period till 3 days after end of second treatment period (day 25 or 32).
Arm/Group | Active | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 9/19 | 6/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=19) | Placebo (N=19)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Blood immunoglobulin E increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram ST segment elevation (Investigations) | 0 (0) | 1 (1)
Low density lipoprotein increased (Investigations) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor seeks publication of all clinical trials in peer-reviewed journals within 18 months after completion or termination of the clinical trial, regardless of whether the findings are positive or negative. If no publication is submitted by the sponsor within these 18 months, the investigator has the right to publish the results from the clinical trial generated by him/herself.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT04853992/Prot_SAP_001.pdf